CLINICAL TRIAL: NCT02245932
Title: The Effect of Resveratrol on Metabolism and Cardiovascular Risk Profile in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Resveratrol In Chronic Obstructive Pulmonary Disease (COPD) Patients (CARMENS-trial)
Acronym: CARMENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Netherlands Asthma Foundation (Other); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 143031; 3.4.12.023 (Other Grant/Funding Number: The Netherlands Lung Foundation)
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2016-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary disease, Chronic Obstructive; Cardiovascular diseases; Metabolism; Resveratrol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases | interventions — Resveratrol; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol supplementation (Experimental): 150 mg of resveratrol for 4 weeks (split over two doses of 75 mg/day)
  Interventions: Dietary Supplement: Resveratrol
- Placebo supplementation (Placebo Comparator): Placebo for 4 weeks (split over two doses per day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — 4 weeks of 150 mg resveratrol (2 times 75mg/day)
  Other Names: resVida (99% pure trans-resveratrol) provided by DSM Nutritional Products, Ltd.
  Arms: Resveratrol supplementation
Dietary Supplement: Placebo — 4 weeks of placebo supplementation (two doses per day)
  Arms: Placebo supplementation

SUMMARY:
The primary objective is to investigate the efficacy of resveratrol on mitochondrial function in patients with COPD. The secondary objective is to investigate the effect of resveratrol on body composition, inflammatory status and mechanistic markers in blood, adipose and muscle tissue as well as a comprehensive assessment of metabolicand physical performance profile known to be affected by resveratrol.

DETAILED DESCRIPTION:
Rationale: Patients with COPD are often chaacterized by disturbed metabolic health affecting physical and cognitive function, which is reflected in altered body composition. current studies in healthy subjects suggest that resveratrol improves metabolic health by enhancing muscle mitochondrial function and adipose tissue morphology.

Study design: Proof-of-concept randomized placebo-controlled double blinded clinical trial of 4 weeks.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects may be confronted with certain inconveniences and risks. Subjects will be asked to wear an accelerometer two times for one week. During the entire study period subjects will visit the MUMC+ 2 times for various non-invasive measurements (questionnaires, anthropometry, and physical function test) as well as some minor invasive procedures (venous blood sampling and muscle and fat biopsies) which can cause a local haematoma afterwards. However, the patients will be informed about their metabolic and cardiovascular health, which we expect to be positively affected by the intervention. In addition, all patients will receive a lifestyle advice tailored to their health status.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* Current or ex-smoker
* Age >18 years

Exclusion Criteria:

* COPD patients planned for pulmonary rehabilitation or who recently participated in a rehabilitation program in the previous 6 months
* Investigator's uncertainty about willingness or ability of the patient to comply with the protocol requirements
* Participation in any other study involving investigational exercise training, nutritional or pharmacological intervention
* Oral glucocorticoid use
* Recent exacerbation (<4 weeks) that required oral steroids and/or hospital admission
* Subject is pregnant, planning to be pregnant during the study period, lactating, or women who consider themselves to be of childbearing potential and who are engaged in an active sex life and are unwilling to commit to the use of an approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation;
* Diabetes mellitus (all types), active cardiovascular disease or a cardiovascular event (such as myocardial infarction, cerebrovascular haemorrhage/infarction) in the previous 6 months, recent major surgery, thyroid dysfunction, hepatic or renal disorders, current malignancy (except for dermal malignancies) or central or obstructive sleep apnea;
* Current alcohol consumption > 20 grams alcohol/day;
* Intake of resveratrol containing dietary supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in mitochondrial function | 0 and 4 weeks
  Assessed by measuring mitochondrial respiration (using the oxygraph) of a muscle biopsy of the quadriceps muscle (vastus lateralis)

SECONDARY OUTCOMES:
Change from baseline in high sensitivity systemic inflammation (CRP) at 4 weeks | 0 and 4 weeks
  High sensitivity C-reactive protein (CRP) as a clinical marker of systemic inflammation via blood sampling.
Change in adipose tissue inflammation | 0 and 4 weeks
  Assessed by adipose tissue biopsy
Change in systematic inflammatory profile | 0 and 4 weeks
  Assessed via blood sampling
Change in lipid profile | 0 and 4 weeks
  Assessed via blood sampling
Change in insulin sensitivity | 0 and 4 weeks
  Assessed by HOMA-IR
Change in body composition | 0 and 4 weeks
  Assessed by:
  * DEXA-scan
  * Anthropometric measurements
Change in quadriceps function | 0 and 4weeks
  Assessed by leg dynamometry (Biodex)
Change in blood pressure | 0 and 4 weeks
  Measured with a hematometer
Change in heart rate | 0 and 4 weeks
  Measured with a hematometer

OTHER OUTCOMES:
Medical history | 0 and 4 weeks
  Medication use
Physical activity | 0 and 4 weeks
  Assessed by:
  * Accelerometry
  * Short Questionnaire to Assess Health (SQUASH)
Severity of dyspnea and COPD | 0 and 4 weeks
  Assessed by:
  * Medical Research Council scale (MRC-scale)
  * COPD assessment test (CAT)
  * Clinical COPD Questionnaire (CCQ)
Sleep pattern | 0 and 4 weeks
  Assess by Pittburgh Sleep Quality Index (PSQI)
Food intake | 0 and 4 weeks
  Assessed by food anamnesis questionnaire
Resveratrol and dihydroresveratrol concentrations | 0 and 4 weeks
  Assessed by blood sampling
Electrocardiogram | 0 and 4 weeks
  Measured with a ECG
Safety parameters | 0 and 4 weeks
  Assessed in blood:
  * Creatinine
  * Urea
  * Sodium
  * Potassium
  * Gamma-GT
  * ALAT
  * ASAT
  * Alkaline Phosphatase
Baseline lung function | 0 weeks
  Assessed by spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Schols, Prof., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Timmers S, Konings E, Bilet L, Houtkooper RH, van de Weijer T, Goossens GH, Hoeks J, van der Krieken S, Ryu D, Kersten S, Moonen-Kornips E, Hesselink MKC, Kunz I, Schrauwen-Hinderling VB, Blaak E, Auwerx J, Schrauwen P. Calorie restriction-like effects of 30 days of resveratrol supplementation on energy metabolism and metabolic profile in obese humans. Cell Metab. 2011 Nov 2;14(5):612-22. doi: 10.1016/j.cmet.2011.10.002. PMID 22055504
- [Background] van den Borst B, Gosker HR, Schols AM. Central fat and peripheral muscle: partners in crime in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 Jan 1;187(1):8-13. doi: 10.1164/rccm.201208-1441OE. No abstract available. PMID 23281350
- [Derived] Beijers RJ, Gosker HR, Sanders KJ, de Theije C, Kelders M, Clarke G, Cryan JF, van den Borst B, Schols AM. Resveratrol and metabolic health in COPD: A proof-of-concept randomized controlled trial. Clin Nutr. 2020 Oct;39(10):2989-2997. doi: 10.1016/j.clnu.2020.01.002. Epub 2020 Jan 13. PMID 31996311